CLINICAL TRIAL: NCT06064201
Title: The Role of Short-chain Fatty Acids (SCFAs) in Regulating Stress Responses, Eating Behavior, and Nutritional State in Anorexia Nervosa: a Randomized Controlled Trial
Brief Title: The Role of Short-chain Fatty Acids in Malnutrition on Stress, Eating Behavior, and Nutritional State
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Elske Vrieze, Professor dr., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: S66404
Record Dates: First submitted 2023-07-28; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Anorexia Nervosa
Keywords: anorexia nervosa; short-chain fatty acids; gut-brain axis; microbiota; stress response; eating behavior; gut microbiome; food choice; Trier Social Stress Test; randomized controlled trial
MeSH Terms: conditions — Anorexia Nervosa; Fractures, Stress; Feeding Behavior | interventions — Fatty Acids, Volatile

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-chain fatty acids (SCFAs) (Experimental): SCFAs will be delivered directly to the colon using pH-dependent colon delivery capsules (CDCs).
  Interventions: Other: Short-chain fatty acids (SCFAs)
- Microcrystalline cellulose (Placebo Comparator): Placebo capsules
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Short-chain fatty acids (SCFAs) — The SCFAs mixture contains acetate, butyrate, and propionate in a ratio of 60:20:20, and the total daily amount of SCFAs is equivalent to the fermentation of 10g of arabinoxylan oligosaccharides. Participants will be asked to consume these capsules spread at four intervals throughout the day. The nursing staff will distribute the capsules to the participants individually, supervise their intake, and monitor adherence by capsule count.
  Arms: Short-chain fatty acids (SCFAs)
Other: Placebo — To serve as a placebo, microcrystalline cellulose will be included in the same type of CDCs.
  Arms: Microcrystalline cellulose

SUMMARY:
This clinical trial aims to test the psychobiological effects of certain substances produced by gut bacteria, known as short-chain fatty acids (SCFAs), in people with anorexia nervosa.

DETAILED DESCRIPTION:
Objective This protocol proposes investigating the effects of short-chain fatty acids (SCFAs), produced by gut bacterial fermentation of dietary fiber, as mediators of microbiota-gut-brain interactions on the acute stress response, eating behavior, and nutritional state in malnourished patients with anorexia nervosa (AN). SCFAs have recently been proposed as crucial mediators of the microbiome's effects on the host. Emerging evidence suggests that SCFAs impact human physiology through various physiological pathways and may regulate stress responses and eating behavior.

Method The investigators will conduct a randomized, triple-blind, placebo-controlled trial in 92 AN patients. Patients will receive either a placebo or a mixture of SCFAs (acetate propionate, butyrate) using colon-delivery capsules (CDCs) for six weeks. This clinical trial is an add-on to the standard inpatient psychotherapeutic program focusing on nutritional rehabilitation.

Hypotheses The investigators hypothesize that colonic SCFAs delivery will modulate neuroendocrine, cardiovascular, and subjective responses to an acute laboratory psychosocial stress task. As secondary outcome measures, the investigators will assess alterations in restrictive eating behavior and nutritional status, as reflected by changes in body mass index (BMI). Additionally, the investigators will explore changes in microbiota composition, gastrointestinal symptoms, eating disorder psychopathology, and related comorbidities.

Discussion The findings of this study can enhance our understanding of how gut microbiota-produced metabolites, particularly SCFAs, impact the stress response and eating behavior of individuals with AN. It has the potential to provide essential insights into the complex interplay between the gut, stress system, and eating behavior and facilitate new therapeutic targets for stress-related psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* Participants are female.
* Participants are at least 16 years of age.
* Participants are Dutch-speaking.
* Participants meet the diagnostic criteria of anorexia nervosa based on the criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5; American Psychiatric Association, 2013). The first time the participant met these criteria was less than seven years ago.
* Participants have a current BMI < 17,5 (kg/m2).
* Participants are on the waiting list for a psychiatric/psychotherapeutic inpatient treatment program with nutritional rehabilitation on the eating disorder ward of the University Psychiatric Hospital Leuven.
* Participants can access a -18°C home freezer for stool storage.

Exclusion Criteria:

* Any medical or psychiatric disorder, which in the Investigator's opinion, might jeopardize the participant's safety or compliance with the protocol.
* Any prior or concomitant treatment(s) that might jeopardize the participant's safety or that would compromise the integrity of the Trial.
* Substance/alcohol/illegal drug abuse or dependence or evidence for chronic uses of sedatives, drugs and/or sleep medication.
* High caffeine intake (> 1000 ml coffee daily or equivalent quantities of other caffeine-containing substances).
* Use of pre- or probiotics within the last month before the start of the study.
* Use of antibiotics within the last three months before the start of the study.
* Pregnancy or intention to become pregnant.
* Previous experience with one of the tasks used in the study.
* Use of antipsychotics
* Use of selective serotonin reuptake inhibitors (SSRIs), oral contraceptives, or other drugs is allowed if patients are on a stable dosage for at least four weeks.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Salivary cortisol response following TSST | Baseline (at hospital admission and before intervention) and post-intervention (following six weeks of intervention)
  Changes in salivary cortisol levels in response to acute laboratory stress (Trier Social Stress Test).
Restrictive food choices during Food Choice Task | Baseline (at hospital admission and before intervention) and post-intervention (following six weeks of intervention)
  Food choices made under stress are measured through the food choice task, focusing on the proportion of high-fat food items chosen over the reference item.
Nutritional status (BMI) | Baseline (at hospital admission and before intervention) and post-intervention (following six weeks of intervention) and at the follow-up visit (12 weeks following the start of the intervention)
  Nutritional status of participants determined by calculating Body Mass Index (BMI) from recurrently measured weight

SECONDARY OUTCOMES:
Neuroendocrine Measures (salivary alpha amylase) | Baseline (at hospital admission and before intervention) and post-intervention (following six weeks of intervention)
  Salivary alpha-amylase (sAA) levels are measured using salivary samples in response to acute laboratory stress (Trier Social Stress Test).
Neuroendocrine Measures (ACTH) | Baseline (at hospital admission and before intervention) and post-intervention (following six weeks of intervention)
  Adrenocorticotropic hormone (ACTH) serum levels are measured in response to acute laboratory stress (Trier Social Stress Test).
Subjective stress in relation to TSST | Baseline (at hospital admission and before intervention) and post-intervention (following six weeks of intervention)
  Participants' subjective subjective stress experience in response to acute laboratory stress is measured using Visual Analog Scales (VAS, scale 0-100), where higher scores indicate higher subjective stress.
Subjective stress appraisal in relation to TSST | Baseline (at hospital admission and before intervention) and post-intervention (following six weeks of intervention)
  The Primary Appraisal and Secondary Appraisal (PASA) scale assesses various stress-related cognitive processes in anticipation of the TSST. The scale comprises four sub-scales: Threat, Challenge, Outcome Expectancy, and Self-efficacy. The first two address issues related to primary appraisal, and the latter two focus on secondary appraisal. Finally, an overall score for perceived stress can also be calculated from PASA by subtracting the secondary appraisal score from that of primary appraisal. Higher scores reflect a more positive anticipatory cognitive stress appraisal.
Subjective anxiety in relation to TSST | Baseline (at hospital admission and before intervention) and post-intervention (following six weeks of intervention)
  Participants' subjective experience of anxiety in response to acute laboratory stress is measured using Visual Analog Scales (VAS, scale 0-100). Higher scores indicate a higher subjective anxiety experience.
Subjective hunger in relation to TSST | Baseline (at hospital admission and before intervention) and post-intervention (following six weeks of intervention)
  Participants' subjective experience of hunger in response to acute laboratory stress is measured using Visual Analog Scales (VAS, scale 0-100). Higher scores indicate higher subjective hunger.
Subjective appetite in relation to TSST | Baseline (at hospital admission and before intervention) and post-intervention (following six weeks of intervention)
  Participants' subjective experience of appetite in response to acute laboratory stress is measured using Visual Analog Scales (VAS, scale 0-100). Higher scores indicate higher subjective appetite.
Heart rate response to acute laboratory stress | Baseline (at hospital admission and before intervention) and post-intervention (following six weeks of intervention)
  Physiological measures to acute laboratory stress: measurement of( autonomic nervous system activity) heart rate response (unit: beats per minute) to acute laboratory stress using EmbracePlus wearable wrist device.
Heart rate variability to acute laboratory stress | Baseline (at hospital admission and before intervention) and post-intervention (following six weeks of intervention)
  Physiological measures to acute laboratory stress: measurement of( autonomic nervous system activity) heart rate variability (unit: milliseconds) to acute laboratory stress using EmbracePlus wearable wrist device.
Electrodermal activity to acute laboratory stress | Baseline (at hospital admission and before intervention) and post-intervention (following six weeks of intervention)
  Physiological measures to acute laboratory stress: measurement of( autonomic nervous system activity) Electrodermal activity (unit: micro siemens) to acute laboratory stress using EmbracePlus wearable wrist device.
Self controlled choices during Food Choice Task | Baseline (at hospital admission and before intervention) and post-intervention (following six weeks of intervention)
  The proportion of self-controlled choices, choosing healthy, less tasty foods or not choosing unhealthy, tasty foods during the food choice task
Eating Disorder Symptoms | Self-reported questionnaires are completed at the baseline visit (at hospital admission and before intervention), three weeks into the intervention, post intervention (following six weeks of intervention) and at the follow-up visit (12 weeks following
  The severity of eating disorder symptoms is evaluated using the Eating Disorder Examination Questionnaire (EDE-Q). The EDE-Q is a 28-item self-report questionnaire adapted from the semi-structured interview, the Eating Disorder Examination (EDE). The questionnaire is designed to assess the range, frequency, and severity of behaviors associated with a diagnosis of an eating disorder. Higher scores indicate more problematic eating behaviors and attitudes.
Restrained, emotional and external eating behaviour | Self-reported questionnaires are completed at the baseline visit (at hospital admission and before intervention), three weeks into the intervention, post intervention (following six weeks of intervention) and at the follow-up visit (12 weeks following
  Restrained, emotional and external eating behaviour is evaluated using the Dutch Eating Behavior Questionnaire (DEBQ). The DEBQ is a 33-item self-report questionnaire to assess three distinct eating behaviors in adults: (1) emotional eating, (2) external eating, and (3) restrained eating. Items on the DEBQ range from 1 (never) to 5 (very often), with higher scores indicating greater endorsement of the eating behavior.
Hedonic hunger | Self-reported questionnaires are completed at the baseline visit (at hospital admission and before intervention), three weeks into the intervention, post intervention (following six weeks of intervention) and at the follow-up visit (12 weeks following
  Hedonic hunger is evaluated using the Power of Food Scale (PFS). The PFS assesses the psychological impact of living in food-abundant environments. It measures appetite for, rather than consumption of, palatable foods, at three levels of food proximity (food available, food present, and food tasted). The PFS consists of 15 items, rated on a 5-point Likert scale, assessing preoccupation with palatable foods across three distinct but related domains (contributing to three separate subscales of the measure).

OTHER OUTCOMES:
Short-chain fatty acid levels | Baseline (at hospital admission and before intervention) and post-intervention (following six weeks of intervention)
  Quantification of serum and stool SCFA
Fecal gut microbiota profile | Baseline (at hospital admission and before intervention) and post-intervention (following six weeks of intervention) and at the follow-up visit (12 weeks following the start of the intervention)
  Assessing gut microbiota profile before and after intervention
Gastrointestinal Symptoms | Self-reported questionnaires are completed at the baseline visit (at hospital admission and before intervention), three weeks into the intervention, post intervention (following six weeks of intervention) and at the follow-up visit (12 weeks following
  Gastrointestinal complaints are scored using combining the results of the Gastrointestinal Symptom Rating Scale (GSRS) and the Rome IV questionnaire for functional gastrointestinal disorders. The GSRS is a disease-specific self-report instrument of 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhea, and Constipation. The GSRS has a seven-point Likert-type scale where 1 represents the absence of troublesome symptoms, and 7 represents very troublesome symptoms.
Physical movement | Baseline (at hospital admission and before intervention) and post-intervention (following six weeks of intervention)
  Using raw accelerometry data (m/s2) and motion intensity detection from the Embraceplus wearable wrist device, physical activity will be measured.
Depressive symptoms | Self-reported questionnaires are completed at the baseline visit (at hospital admission and before intervention), three weeks into the intervention, post intervention (following six weeks of intervention) and at the follow-up visit (12 weeks following
  The DASS is a set of three self-report scales designed to measure the negative emotional states of depression, anxiety, and stress. Each of the three DASS scales contains 14 items, divided into subscales of 2-5 items with similar content.
Positive and negative affect | Self-reported questionnaires are completed at the baseline visit (at hospital admission and before intervention), three weeks into the intervention, post intervention (following six weeks of intervention) and at the follow-up visit (12 weeks following
  The PANAS consists of two 10-item mood scales and was developed to provide brief measures of negative affect (NA) and positive affect (PA). Respondents are asked to rate the extent to which they have experienced each particular emotion within a specified time period, on a 5-point scale. The scale points are: 1 'very slightly or not at all', 2 'a little', 3 'moderately', 4 'quite a bit', and 5 'very much'.
Percieved stress | Self-reported questionnaires are completed at the baseline visit (at hospital admission and before intervention), three weeks into the intervention, post intervention (following six weeks of intervention) and at the follow-up visit (12 weeks following
  The Perceived Stress Scale (PSS) is a 10-item instrument designed to measure the degree to which situations in one's life are appraised as stressful. It provides a tool for examining issues about the role of appraised stress levels in the etiology of disease and behavioral disorders. The scale is designed to ask the respondent to rate the frequency of his/her feelings and thoughts related to events and situations that occurred over a selected timeframe. Notably, high PSS scores correlate with higher stress biomarkers, such as cortisol.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ/KU Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication will be made available to other researchers with all identifying information removed.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will become available upon publication with no time limitations.

REFERENCES:
- [Derived] Quagebeur R, Dalile B, Raes J, Van Oudenhove L, Verbeke K, Vrieze E. The role of short-chain fatty acids (SCFAs) in regulating stress responses, eating behavior, and nutritional state in anorexia nervosa: protocol for a randomized controlled trial. J Eat Disord. 2023 Oct 26;11(1):191. doi: 10.1186/s40337-023-00917-6. PMID 37884972